CLINICAL TRIAL: NCT02651116
Title: A PLACEBO-CONTROLLED, DOUBLE-BLIND, RANDOMIZED, PARALLEL GROUP PILOT STUDY TO EVALUATE THE EFFICACY OF DEXTROMETHORPHAN HYDROBROMIDE ON ACUTE COUGH IN A PEDIATRIC POPULATION
Brief Title: Dextromethorphan Pediatric Acute Cough Study
Acronym: CHPA DXM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was prematurely discontinued due to slow enrollment during the 2019/2020 cold season. No safety or efficacy concerns led to the decision to terminate
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A6531002; CHPA DXM (Other: Alias Study Number)
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Cough
Keywords: cough, acute cough, pediatric, Dextromethorphan Hydrobromide, antitussive, ambulatory cough recording device
MeSH Terms: conditions — Cough | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dextromethorphan Hydrobromide (Experimental): 15 mg/ 10 mL: 10 mL of Dextromethorphan Hydrobromide
  Interventions: Drug: Dextromethorphan Hydrobromide; Device: Cough recording device
- Placebo (Placebo Comparator): 10 mL of Placebo
  Interventions: Drug: Placebo; Device: Cough recording device

INTERVENTIONS:
Drug: Dextromethorphan Hydrobromide — 15 mg/ 10 mL: 10 mL of Dextromethorphan Hydrobromide
  Other Names: DXM
  Arms: Dextromethorphan Hydrobromide
Drug: Placebo — 10 mL Placebo
  Arms: Placebo
Device: Cough recording device — FDA approved device validated for use in adults and children
  Other Names: VitaloJAK

SUMMARY:
This is a placebo-controlled, double-blind, randomized, parallel group pilot study in approximately 150 subjects to evaluate the efficacy of dextromethorphan hydrobromide (DXM) on acute cough in a pediatric population. Subjects will be otherwise healthy males and females aged 6-11 inclusive who are experiencing acute cough as a symptom of common cold or upper respiratory tract infection. Subjects must have had onset of symptoms within 3 days of screening and qualify based on physical exam and symptom questionnaire. Eligible subjects will be given a single-blind placebo, and fitted with a cough counting device for a 2 hour run-in period. Qualifying subjects will be stratified by age and then randomized to either DXM or placebo in a 1:1 ratio and fitted with the cough recording device for the first 24 hours of treatment. Subjects will receive approximately 9 doses of investigational product over the course of the 4 day study and will complete patient reported outcome questions before the morning and afternoon doses. Subjects will return to the study site on Day 2 to remove the cough recorder and on Day 4 (+ 2 days) to complete the final visit. A review of any reported adverse events will also be completed.

DETAILED DESCRIPTION:
This is a placebo-controlled, double-blind, randomized, parallel group pilot study in approximately 150 subjects to evaluate the efficacy of dextromethorphan hydrobromide DXM) on acute cough in a pediatric population. Subjects will be otherwise healthy males and females aged 6-11 inclusive who are experiencing acute cough as a symptom of common cold or upper respiratory tract infection. Subjects must have had onset of symptoms within 3 days of screening and qualify based on physical exam and symptom questionnaire. Eligible subjects will be given a single-blind placebo, and fitted with a cough counting device for a 2 hour run-in period. Qualifying subjects will be stratified by age and then randomized to either DXM or placebo in a 1:1 ratio and fitted with the cough recording device for the first 24 hours of treatment. Subjects will receive approximately 9 doses of investigational product over the course of the 4 day study and will complete patient reported outcome questions before the morning and afternoon doses. Subjects will return to the study site on Day 2 to remove the cough recorder and Day 4 (+2 days) to complete the final visit. A review of any reported adverse events will also be completed. Validated Patient Reported Outcomes (PRO) used in the study include morning cough assessment, afternoon cough assessment, Child Global Question, and Child Cold Symptom Checklist

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy male or female children/adolescents ages 6 to 11 years, inclusive.
* Subject has an acute cough and other symptoms consistent with a common cold/acute upper respiratory tract infection (URTI) diagnosis as deemed by the investigator or qualified designee based on findings from medical history review, full physical examination and vital signs.
* The onset of symptoms must be no more than 3 days prior to Visit 1, as determined by the subject or parent/legally acceptable representative.
* Qualifying response on the Child Cold Symptom Checklist.
* Parent/legally acceptable representative, and subject agrees the subject will not use any other cough or cold treatments during the study.

Exclusion Criteria:

* A subchronic, or chronic cough due to any condition other than an URTI or common cold as established by the investigator, nurse practitioner, or physician's assistant, in accordance with the American College of Chest Physicians' (ACCP) Guidelines for Diagnosis and Management of Cough. Special attention should be paid to highly prevalent conditions commonly presenting with cough such as asthma, rhinitis, or gastroesophageal reflux disease (GERD).
* Symptoms of runny nose, stuffy nose, sore throat, or sneezing due to any condition other than URTI or common cold (eg, seasonal or perennial allergic rhinitis, sinusitis, strep throat, vasomotor rhinitis, etc.) as established by the investigator.
* An acute cough that occurs with excessive phlegm (mucus) or is chronic such as occurs with smoking, asthma, bronchitis, allergies, or a gastroesophageal condition (eg, acid reflux and GERD) or history of such a cough.
* Clinical features of a complication of the common cold during the physical examination at screening (eg, otitis media, sinusitis, or pneumonia) with or without the need for systematic antibiotics.
* Pneumonia (active or with a symptom-free period of <30 days), asthma (active or with a symptom-free period of <1 year), or other significant pulmonary diseases.
* Fever greater than 39ºC (102ºF oral temperature) at the time of screening if, in the judgment of the investigator, the individual is too ill to participate in the study or the fever is due to reasons other than URTI.
* Signs of dehydration (as may be due to vomiting, diarrhea, or lack of fluid intake) during the physical examination at screening.
* Diabetes or hypoglycemic disorders.
* Known contraindications to the investigational product or acetaminophen (APAP).
* Sitting blood pressure reading at or above the limits as documented in the protocol.
* Obstructive sleep apnea caused by enlarged tonsils and adenoids, low muscle tone, or allergies.
* History of known or suspected allergy or hypersensitivity to dextromethorphan (DXM) or APAP, or any of the non medicinal ingredients contained in the single-blind confection, double-blind investigational products, or APAP.
* History of taking any of the specified prohibited medications or products within the corresponding washout periods prior to taking the first dose of investigational product.
* History of taking a medication that is sedating within the past 24 hours prior to screening (eg sedatives, hypnotics, tranquilizers, anticonvulsants, benzodiazepines, and clonidine).
* Subject has a sibling contemporaneously participating in this study.

Randomization Criteria:

* Subjects must complete the 2 hour ambulatory cough counting baseline run-in recording period and must return to the study site for randomization at least 2 hours after the recording started.
* Subjects whose equipment failed, preventing collection of cough count data for at least 2 hours during the Baseline Run-in Period, or those who took off the device during this period will be excluded from further study participation.
* Subjects who do not return to the study site (before 3:30 pm) in time for the afternoon dose will not be randomized.
* Qualifying response on Child Global Question

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (18):
  - Avail Clinical Research, LLC, DeLand, Florida
  - Clinical Associates of Orlando LLC, Orlando, Florida
  - Elite Clinical Trials LLLP, Blackfoot, Idaho
  - Advanced Clinical Research, Meridian, Idaho
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - All Children Pediatrics, Louisville, Kentucky
  - Bluegrass Clinical Research, Inc, Louisville, Kentucky
  - MedPharmics, LLC, Metairie, Louisiana
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Meridian Clinical Research LLC, Omaha, Nebraska
  - Rapid Medical Research, Inc, Cleveland, Ohio
  - Coastal Pediatric Associates, Charleston, South Carolina
  - Coastal Pediatric Associates, Mt. Pleasant, South Carolina
  - Carolina Ear, Nose & Throat Clinic/CENTRI Inc., Orangeburg, South Carolina
  - Meridian Clinical Research, LLC, Dakota Dunes, South Dakota
  - Texas Health Care, PLLC, Fort Worth, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Advanced Clinical Research, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6531002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in the United States from 25 February 2016 to 19 March 2020.
Pre-assignment Details: There was a run-in period of 2 hours where participants were administered 10 milliliter (mL) of non-medicinal liquid oral confection for once, and fitted with cough counting device VitaloJAKTM. Eligible participants who completed run-in period, were qualified for randomization to either dextromethorphan hydrobromide (DXM HBr) or placebo in a 4 day treatment period.
Groups:
- Dextromethorphan Hydrobromide: Participants were randomized to receive 9 doses of DXM HBr (15 milligram [mg] per 10 mL) over the course of 4 day study treatment and were fitted with the cough recording device VitaloJAKTM for the first 24 hours of treatment. On Day 1, participants received a single 10 mL oral dose of DXM HBr syrup each in afternoon and evening. On Day 2 and 3, participants received a single 10 mL oral dose of DXM HBr syrup each in morning, afternoon and evening. On Day 4, participants received a single 10 mL oral dose of DXM HBr syrup in morning. Participants were followed up for 14 days after last dose of study medication.
- Placebo: Participants were randomized to receive 9 doses of placebo matched to 15 mg/10 mL DXM HBr over the course of 4 day study treatment and were fitted with the cough recording device VitaloJAKTM for the first 24 hours of treatment. On Day 1, participants received a single 10 mL oral dose of placebo syrup each in afternoon and evening. On Day 2 and 3, participants received a single 10 mL oral dose of placebo syrup each in morning, afternoon and evening. On Day 4, participants received a single 10 mL oral dose of placebo syrup in morning. Participants were followed up for 14 days after last dose of study medication.
Period: Overall Study
Arm/Group | Dextromethorphan Hydrobromide | Placebo
Started | 68 | 63
Treated | 68 | 63
Completed | 67 | 62
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — No Longer Willing To Participate In Study | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received the study drug.
Groups:
- Dextromethorphan Hydrobromide: Participants were randomized to receive 9 doses of DXM HBr (15 mg/10 mL) over the course of 4 day study treatment and were fitted with the cough recording device VitaloJAKTM for the first 24 hours of treatment. On Day 1, participants received a single 10 mL oral dose of DXM HBr syrup each in afternoon and evening. On Day 2 and 3, participants received a single 10 mL oral dose of DXM HBr syrup each in morning, afternoon and evening. On Day 4, participants received a single 10 mL oral dose of DXM HBr syrup in morning. Participants were followed up for 14 days after last dose of study medication.
- Total: Total of all reporting groups
Arm/Group | Dextromethorphan Hydrobromide | Placebo | Total
Number analyzed (Participants) | 68 | 63 | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.3 (1.57) | 8.0 (1.73) | 8.2 (1.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 67
  Male | 33 | 31 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 64 | 56 | 120
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 22 | 46
  White | 40 | 39 | 79
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean of Total Cough Counts: Over 24 Hours Post-First Dose on Day 1
Description: Total cough count was collected by the cough recording device VitaloJAKTM in an ambulatory setting. The VitaloJAKTM device recorded continuous digital audio obtained through both a lapel microphone clipped to the participant's clothing at the neck or upper chest level, and a chest wall sensor attached to the participant's chest at the top of the sternum. Data was captured on a data card and the vitalograph analyst evaluated cough counts.
Time Frame: Over for 24 hours post-first dose on Day 1
Population: The full analysis set included all participants who were randomized, took Dose 1, had a valid baseline cough count assessment, and provided any post-dosing efficacy data.
Measure: Mean (Standard Deviation); unit: cough counts
Arm/Group | Dextromethorphan Hydrobromide | Placebo
Number analyzed (Participants) | 67 | 61
cough counts | 457.1 (367.21) [lower limit 367.21] | 676.8 (814.33) [lower limit 814.33]
Statistical Analysis 1: Comparison: Dextromethorphan Hydrobromide vs Placebo; Estimated rate ratio (ratio of rate of cough counts per 24 hours for DXM HBr to placebo), and corresponding 95% confidence interval (CI) for DXM HBr versus placebo was obtained from negative binomial model with treatment, study site (pooled), age group, and log-transformed baseline average cough count per hour as factors, with logarithm of the time over which the cough count was evaluated as the offset parameter; Test type: Superiority; p = 0.0449, Negative Binomial Regression — P-Value less than or equal to (<=) 0.05 level was considered significantly better and P-Value lying between 0.05 less than (<) p<=0.1 level was considered marginally significantly better; Rate Ratio = 0.7899, 95% CI 2-sided [0.6273 to 0.9947], Standard Error of Mean 0.0929
Statistical Analysis 2: Comparison: Dextromethorphan Hydrobromide vs Placebo; P-value was obtained from the negative binomial model with treatment, study site (pooled), age group, log-transformed baseline average cough count per hour (based on Baseline Run-in Period) as factors, with interaction term of treatment by age group, and logarithm of the time over which the cough count was evaluated as the offset parameter; Test type: Superiority; p = 0.6293, Negative Binomial Regression — P-value is for interaction term of treatment by age group. P-value <=0.10 was considered significant for interaction terms

2. Secondary Outcome: Mean of Total Cough Counts: Between Dose 1 to Dose 2 on Day 1
Description: as for outcome 1
Time Frame: Between Dose 1 to Dose 2 on Day 1
Population: The full analysis set included all participants who were randomized, took Dose 1, had a valid baseline cough count assessment, and provided any post-dosing efficacy data. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cough counts
Arm/Group | Dextromethorphan Hydrobromide | Placebo
Number analyzed (Participants) | 66 | 61
cough counts | 32.73 (30.597) [lower limit 30.597] | 47.03 (57.729) [lower limit 57.729]
Statistical Analysis 1: Comparison: Dextromethorphan Hydrobromide vs Placebo; Estimated rate ratio (ratio of rate of cough counts per specified duration for DXM HBr to placebo, used in evaluation of this outcome measure), and corresponding 95% CI for DXM HBr versus placebo was obtained from negative binomial model with treatment, study site (pooled), age group, and log-transformed baseline average cough count per hour as factors, with logarithm of the time over which the cough count was evaluated as the offset parameter; Test type: Superiority; p = 0.0552, Negative Binomial Regression — P-Value <=0.05 level was considered significantly better and P-Value lying between 0.05<p<=0.1 level was considered marginally significantly better; Rate Ratio = 0.8048, 95% CI 2-sided [0.6446 to 1.0049], Standard Error of Mean 0.0912

3. Secondary Outcome: Mean of Total Cough Counts: Between Dose 2 on Day 1 to Dose 3 on Day 2
Description: as for outcome 1
Time Frame: Between Dose 2 on Day 1 to Dose 3 on Day 2 (second dose of Day 1 to first dose of Day 2)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cough counts
Arm/Group | Dextromethorphan Hydrobromide | Placebo
Number analyzed (Participants) | 65 | 61
cough counts | 9.70 (8.877) [lower limit 8.877] | 11.44 (13.193) [lower limit 13.193]
Statistical Analysis 1: Comparison: Dextromethorphan Hydrobromide vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.7684, Negative Binomial Regression — [p-value comment as in outcome 2, analysis 1]; Rate Ratio = 0.9551, 95% CI 2-sided [0.7032 to 1.2971], Standard Error of Mean 0.1491

4. Secondary Outcome: Mean of Total Cough Counts: Between Dose 3 to Dose 4 on Day 2
Description: as for outcome 1
Time Frame: Between Dose 3 to Dose 4 on Day 2 (between first and second dose of Day 2)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cough counts
Arm/Group | Dextromethorphan Hydrobromide | Placebo
Number analyzed (Participants) | 65 | 60
cough counts | 19.32 (16.752) [lower limit 16.752] | 33.62 (47.709) [lower limit 47.709]
Statistical Analysis 1: Comparison: Dextromethorphan Hydrobromide vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0220, Negative Binomial Regression — [p-value comment as in outcome 2, analysis 1]; Rate Ratio = 0.7014, 95% CI 2-sided [0.5178 to 0.9500], Standard Error of Mean 0.1086

5. Secondary Outcome: Mean of Total Cough Counts: Between Dose 1 to Dose 2 on Day 1, and Between Dose 3 to Dose 4 on Day 2
Description: Total cough count was collected by the cough recording device VitaloJAKTM in an ambulatory setting. The VitaloJAKTM device recorded continuous digital audio obtained through both a lapel microphone clipped to the participant's clothing at the neck or upper chest level, and a chest wall sensor attached to the participant's chest at the top of the sternum. Data was captured on a data card and the vitalograph analyst evaluated cough counts. In this outcome measure, as planned combined data is reported for first dosing interval (Dose 1 to Dose 2) on Day 1 and first dosing interval (Dose 3 to Dose 4) on Day 2.
Time Frame: Duration between Dose 1 to Dose 2 on Day 1 (between first and second dose of Day 1) plus duration between Dose 3 to Dose 4 on Day 2 (between first and second dose of Day 2)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cough counts
Arm/Group | Dextromethorphan Hydrobromide | Placebo
Number analyzed (Participants) | 66 | 61
cough counts | 26.13 (21.498) [lower limit 21.498] | 40.39 (49.896) [lower limit 49.896]
Statistical Analysis 1: Comparison: Dextromethorphan Hydrobromide vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0098, Negative Binomial Regression — [p-value comment as in outcome 2, analysis 1]; Rate Ratio = 0.7454, 95% CI 2-sided [0.5964 to 0.9316], Standard Error of Mean 0.0848

6. Secondary Outcome: Mean of Total Cough Time Accumulated Over a 24-Hour Period Post-First Dose on Day 1
Description: Time (in seconds) accumulated over a 24-hour period when cough events occurred was collected by the cough recording device VitaloJAKTM in an ambulatory setting. The VitaloJAKTM device recorded continuous digital audio obtained through both a lapel microphone clipped to the participant's clothing at the neck or upper chest level, and a chest wall sensor attached to the participant's chest at the top of the sternum. Data was captured on a data card and the vitalograph analyst evaluated total cough time accumulated.
Time Frame: Over for 24 hours post-first dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Dextromethorphan Hydrobromide | Placebo
Number analyzed (Participants) | 67 | 61
seconds | 350.5 (268.95) [lower limit 268.95] | 502.7 (566.57) [lower limit 566.57]
Statistical Analysis 1: Comparison: Dextromethorphan Hydrobromide vs Placebo; Analysis of covariance (ANCOVA) model contained treatment, study site (pooled), log-transformed baseline cough time and age group terms as factors; Test type: Superiority; p = 0.0977, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Difference in least squares mean = -0.2210, 95% CI 2-sided [-0.4831 to 0.0411], Standard Error of Mean 0.1324

7. Other Pre Specified Outcome: Change From Baseline in Morning Cough Frequency Assessed in Morning at Day 2, 3, and 4
Description: Participants on specified time points were asked to respond to the following question: "from when you woke up this morning until now, how much have you been coughing", on a 5-point scale: 0= not at all, 1= a tiny bit, 2= a little, 3= some and 4= a lot. Higher scores indicated higher frequency of cough in morning time.
Time Frame: Baseline (morning screening visit on Day 1); Within 30 minutes of waking, before morning dose on Days 2, 3, and 4
Population: The full analysis set included all participants who were randomized, took Dose 1, had a valid baseline cough count assessment, and provided any post-dosing efficacy data. Here 'number analyzed' signifies participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dextromethorphan Hydrobromide | Placebo
Number analyzed (Participants) | 67 | 61
units on a scale
  Baseline | 3.4 (0.65) | 3.3 (0.63)
  Change at Day 2: number analyzed (Participants) | 66 | 61
  Change at Day 2 | -1.2 (1.30) | -0.7 (1.15)
  Change at Day 3: number analyzed (Participants) | 66 | 60
  Change at Day 3 | -1.5 (1.15) | -1.1 (1.38)
  Change at Day 4: number analyzed (Participants) | 66 | 60
  Change at Day 4 | -2.0 (1.20) | -1.8 (1.40)
Statistical Analysis 1: Comparison: Dextromethorphan Hydrobromide vs Placebo; Analysis of variance (ANOVA) model contained treatment, study site (pooled), the corresponding morning baseline cough frequency by participant, and age group included in the model. The statistical analysis was performed on the composite for all categories; Test type: Superiority; p = 0.0191, ANOVA — [p-value comment as in outcome 2, analysis 1]; Difference in least squares mean = -0.2881, 95% CI 2-sided [-0.5287 to -0.0475], Standard Error of Mean 0.1224
Statistical Analysis 2: Comparison: Dextromethorphan Hydrobromide vs Placebo; ANOVA model contained treatment, study site (pooled), screening assessment by participant, interaction of treatment by age group and age group included in the model; Test type: Superiority; p = 0.8355, ANOVA — [p-value comment as in outcome 1, analysis 2]

8. Other Pre Specified Outcome: Change From Baseline in Morning Cough Severity Assessed in Morning at Day 2, 3, and 4
Description: Participants on specified time points were asked to respond to the following question: "how bad is your cough this morning", on a 5-point scale: 0= no cough, 1= a tiny bit bad, 2= a little bad, 3= bad and 4= very bad. Higher scores indicated more severe cough in morning time.
Time Frame: Baseline (morning screening visit on Day 1); Within 30 minutes of waking, before morning dose on Days 2, 3, and 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dextromethorphan Hydrobromide | Placebo
Number analyzed (Participants) | 67 | 61
units on a scale
  Baseline | 3.1 (0.54) | 3.1 (0.60)
  Change at Day 2: number analyzed (Participants) | 66 | 61
  Change at Day 2 | -1.1 (0.89) | -0.6 (1.19)
  Change at Day 3: number analyzed (Participants) | 66 | 60
  Change at Day 3 | -1.4 (0.96) | -1.3 (1.22)
  Change at Day 4: number analyzed (Participants) | 66 | 60
  Change at Day 4 | -1.9 (1.10) | -1.8 (1.15)
Statistical Analysis 1: Comparison: Dextromethorphan Hydrobromide vs Placebo; ANOVA model contained treatment, study site (pooled), the corresponding morning baseline cough severity by participant, and age group included in the model. The statistical analysis was performed on the composite for all categories; Test type: Superiority; p = 0.0049, ANOVA — [p-value comment as in outcome 2, analysis 1]; Difference in least squares mean = -0.3128, 95% CI 2-sided [-0.5299 to -0.0956], Standard Error of Mean 0.1104
Statistical Analysis 2: Comparison: Dextromethorphan Hydrobromide vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.8413, ANOVA — [p-value comment as in outcome 1, analysis 2]

9. Other Pre Specified Outcome: Change From Baseline in Impact of Cough on Sleep Assessed in Morning at Day 2, 3, and 4
Description: Participants on specified time points were asked to respond to the following question: "last night in bed, how much did your cough keep you awake", on a 5-point scale: 0= not at all, 1= a tiny bit, 2= a little, 3= some and 4= a lot. Higher scores indicated worse impact of cough on sleep.
Time Frame: Baseline (morning screening visit on Day 1); Within 30 minutes of waking, before morning dose on Days 2, 3, and 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dextromethorphan Hydrobromide | Placebo
Number analyzed (Participants) | 67 | 61
units on a scale
  Baseline | 2.8 (1.15) | 3.0 (1.19)
  Change at Day 2: number analyzed (Participants) | 66 | 61
  Change at Day 2 | -0.8 (1.56) | -0.7 (1.45)
  Change at Day 3: number analyzed (Participants) | 66 | 60
  Change at Day 3 | -1.3 (1.59) | -1.4 (1.67)
  Change at Day 4: number analyzed (Participants) | 66 | 60
  Change at Day 4 | -1.8 (1.57) | -1.9 (1.74)
Statistical Analysis 1: Comparison: Dextromethorphan Hydrobromide vs Placebo; ANOVA model contained treatment, study site (pooled), the corresponding morning baseline impact on sleep by participant, and age group included in the model. The statistical analysis was performed on the composite for all categories; Test type: Superiority; p = 0.2679, ANOVA — [p-value comment as in outcome 2, analysis 1]; Difference in least squares mean = -0.1483, 95% CI 2-sided [-0.4112 to 0.1146], Standard Error of Mean 0.1337
Statistical Analysis 2: Comparison: Dextromethorphan Hydrobromide vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.2882, ANOVA — [p-value comment as in outcome 1, analysis 2]

10. Other Pre Specified Outcome: Change From Baseline in Afternoon Cough Frequency Assessed at Afternoon on Day 2, 3, and 4
Description: Participants on specified time points were asked to respond to the following question: "how much have you been coughing this afternoon" on a 5-point scale: 0= not at all, 1= a tiny bit, 2= a little, 3= some and 4= a lot. Higher scores indicated higher frequency of cough in afternoon time.
Time Frame: Baseline (afternoon visit on Day 1 before first dose); Before the afternoon dose on Day 2, and 3; Anytime in afternoon of Day 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dextromethorphan Hydrobromide | Placebo
Number analyzed (Participants) | 67 | 61
units on a scale
  Baseline | 3.2 (0.80) | 3.4 (0.73)
  Change at Day 2: number analyzed (Participants) | 66 | 61
  Change at Day 2 | -0.7 (1.25) | -0.6 (1.06)
  Change at Day 3: number analyzed (Participants) | 66 | 60
  Change at Day 3 | -1.5 (1.30) | -1.4 (1.27)
  Change at Day 4: number analyzed (Participants) | 63 | 58
  Change at Day 4 | -1.9 (1.22) | -1.8 (1.41)
Statistical Analysis 1: Comparison: Dextromethorphan Hydrobromide vs Placebo; ANOVA model contained treatment, study site (pooled), the corresponding afternoon baseline cough frequency by participant, and age group included in the model. The statistical analysis was performed on the composite for all categories; Test type: Superiority; p = 0.0242, ANOVA — [p-value comment as in outcome 2, analysis 1]; Difference in least squares mean = -0.2812, 95% CI 2-sided [-0.5255 to -0.0369], Standard Error of Mean 0.1242
Statistical Analysis 2: Comparison: Dextromethorphan Hydrobromide vs Placebo; ANOVA model contained treatment, study site (pooled), afternoon baseline assessment by participant, interaction of treatment by age group and age group included in the model; Test type: Superiority; p = 0.2892, ANOVA — [p-value comment as in outcome 1, analysis 2]

11. Other Pre Specified Outcome: Change From Baseline in Afternoon Cough Severity Assessed at Afternoon on Day 2, 3, and 4
Description: Participants on specified time points were asked to respond to the following question: "how bad is your cough this afternoon" on a 5-point scale: 0= no cough, 1= a tiny bit bad, 2= a little bad, 3= bad and 4= very bad. Higher scores indicated more severe cough in afternoon time.
Time Frame: as for outcome 10
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dextromethorphan Hydrobromide | Placebo
Number analyzed (Participants) | 67 | 61
units on a scale
  Baseline | 2.8 (0.83) | 3.1 (0.84)
  Change at Day 2: number analyzed (Participants) | 66 | 61
  Change at Day 2 | -0.7 (1.16) | -0.6 (0.98)
  Change at Day 3: number analyzed (Participants) | 66 | 60
  Change at Day 3 | -1.4 (1.15) | -1.4 (1.24)
  Change at Day 4: number analyzed (Participants) | 63 | 58
  Change at Day 4 | -1.7 (1.08) | -1.6 (1.45)
Statistical Analysis 1: Comparison: Dextromethorphan Hydrobromide vs Placebo; ANOVA model contained treatment, study site (pooled), the corresponding afternoon baseline cough severity by participant, and age group included in the model. The statistical analysis was performed on the composite for all categories; Test type: Superiority; p = 0.0063, ANOVA — [p-value comment as in outcome 2, analysis 1]; Difference in least squares mean = -0.3014, 95% CI 2-sided [-0.5170 to -0.0858], Standard Error of Mean 0.1096
Statistical Analysis 2: Comparison: Dextromethorphan Hydrobromide vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p = 0.3268, ANOVA — [p-value comment as in outcome 1, analysis 2]

12. Other Pre Specified Outcome: Change From Baseline in Child Global Question Assessed at Afternoon on Day 2, 3, and 4
Description: Participants on specified time points were asked to respond to the following question: "how bad is your cold today", on a 5-point scale; 0= no cold, 1= a tiny bit bad, 2= a little bad, 3= bad, and 4= very bad. Higher scores indicated worse cold.
Time Frame: as for outcome 10
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dextromethorphan Hydrobromide | Placebo
Number analyzed (Participants) | 67 | 61
units on a scale
  Baseline | 3.2 (0.42) | 3.3 (0.46)
  Change at Day 2: number analyzed (Participants) | 66 | 61
  Change at Day 2 | -1.1 (1.02) | -0.9 (1.01)
  Change at Day 3: number analyzed (Participants) | 66 | 60
  Change at Day 3 | -1.6 (0.93) | -1.6 (1.13)
  Change at Day 4: number analyzed (Participants) | 63 | 58
  Change at Day 4 | -2.1 (0.87) | -1.7 (1.26)
Statistical Analysis 1: Comparison: Dextromethorphan Hydrobromide vs Placebo; ANOVA model with treatment, study site (pooled), the baseline assessment in child global question cold assessment by participant and age group included in the model. The statistical analysis was performed on the composite for all categories; Test type: Superiority; p = 0.0247, ANOVA — [p-value comment as in outcome 2, analysis 1]; Difference in least squares mean = -0.2535, 95% CI 2-sided [-0.4745 to -0.0325], Standard Error of Mean 0.1124
Statistical Analysis 2: Comparison: Dextromethorphan Hydrobromide vs Placebo; ANOVA model with treatment, study site (pooled), baseline assessment by participant, interaction of treatment by age group and age group included in the model; Test type: Superiority; p = 0.4093, ANOVA — [p-value comment as in outcome 1, analysis 2]

13. Other Pre Specified Outcome: Pediatric Global Assessment of Satisfaction With Study Medication: By Participant, and Caregiver
Description: Participants at the end of the study were asked to respond to the following question: "How would you rate the study medication for taking away your cough?" on a 7-point scale: 0= excellent, 1= very good, 2= good, 3= fair, 4= poor, 5= very poor, and 6= terrible. Higher scores indicated poorer satisfaction with study medication. Within 20 minutes after participants completed the assessment parents/legally acceptable representative were asked to respond to the question: "How would you rate the study medication for taking away your child's cough?" on a 7-point scale: 0= excellent, 1= very good, 2= good, 3= fair, 4= poor, 5= very poor, and 6= terrible. Higher scores indicated poorer satisfaction with study medication.
Time Frame: For participants: at the end of the study on Day 4; For parents/legally acceptable representatives: within 20 minutes after participant completed assessment at the end of the study on Day 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dextromethorphan Hydrobromide | Placebo
Number analyzed (Participants) | 66 | 61
units on a scale
  By Participant: | 1.7 (1.20) | 1.6 (1.26)
  By Caregiver: | 1.8 (1.07) | 1.9 (1.16)
Statistical Analysis 1: Comparison: Dextromethorphan Hydrobromide vs Placebo; Participant: ANOVA model with treatment, study site (pooled), and age group included in the model; Test type: Superiority; p = 0.5652, ANOVA — [p-value comment as in outcome 2, analysis 1]; Difference in least squares mean = 0.1266, 95% CI 2-sided [-0.3081 to 0.5614], Standard Error of Mean 0.2196
Statistical Analysis 2: Comparison: Dextromethorphan Hydrobromide vs Placebo; Caregiver: ANOVA model with treatment, study site (pooled), and age group included in the model; Test type: Superiority; p = 0.4914, ANOVA — [p-value comment as in outcome 2, analysis 1]; Difference in least squares mean = -0.1368, 95% CI 2-sided [-0.5292 to 0.2556], Standard Error of Mean 0.1982
Statistical Analysis 3: Comparison: Dextromethorphan Hydrobromide vs Placebo; Participant: ANOVA model with treatment, study site (pooled), interaction of treatment by age group and age group included in the model; Test type: Superiority; p = 0.1029, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Dextromethorphan Hydrobromide vs Placebo; Caregiver: ANOVA model with treatment, study site (pooled), interaction of treatment by age group and age group included in the model; Test type: Superiority; p = 0.4736, ANOVA — [p-value comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: Day 1 up to 14 days after last dose of study medication (up to 18 days)
Description: Same event may appear as Adverse Event and Serious Adverse Events, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety was evaluated on all participants who received the study drug.
Arm/Group | Dextromethorphan Hydrobromide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/63
Other Adverse Events (participants affected / at risk) | 13/68 | 16/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dextromethorphan Hydrobromide (N=68) | Placebo (N=63)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 2
Otitis media acute (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Headache (Nervous system disorders) | 1 | 3
Dennie-Morgan fold (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal turbinate abnormality (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT02651116/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT02651116/SAP_001.pdf